CLINICAL TRIAL: NCT03794609
Title: An International, Prospective Registry Investigating the Natural History of Participants With Achondroplasia
Brief Title: Observational Study Investigating Clinical & Anthropometric Characteristics of Children With Achondroplasia.
Status: Terminated | Type: Observational
Why Stopped: The study was terminated on 18th November 2022. The decision to terminate the trial was not based on any safety and/or efficacy concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: TA46-002; C4181001 (Other: Alias Study Number)
Record Dates: First submitted 2018-11-19; First posted 2019-01-07 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-07

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a registry study in children with achondroplasia, age 0-10 years, to be conducted at multiple clinical centers in several countries. Information collected will include in anthropometric characteristics, related symptoms, tests, & treatments

Children's information will be collected in the registry for a maximum of 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent is obtained from the children's parent(s) / legal guardian(s) before any study-related activity is carried out
2. The child is able to provide written informed assent, where this is required according to national legislation, before any study related activity is carried out
3. The child has been diagnosed as having achondroplasia documented by clinical diagnosis
4. The child is between 0 years and 10 years of age, inclusive, on the date of consent / assent
5. The investigator has considered the family and prospective participating child being able to comply with the study procedures

Exclusion Criteria:

1. The child has a diagnosis of hypochondroplasia or any short stature condition other than achondroplasia (eg, spondyloepiphyseal dysplasia congenital [SEDC], pseudoachondroplasia, trisomy 21)
2. The child has any medical condition that may impact growth or where the treatment is known to impact growth, such as but not limited to hypothyroidism or hyperthyroidism, insulin-requiring diabetes mellitus, autoimmune inflammatory disease (including celiac disease, systemic lupus erythematosus [SLE], juvenile dermatomyositis, scleroderma, and others), autonomic neuropathy, or inflammatory bowel disease
3. Treatment in the previous 12 months prior to consent and assent with growth hormone, insulin-like growth factor 1 (IGF-1), anabolic steroids, or any other drug expected to affect growth velocity
4. Any surgery that affects the growth plate of the long bones that is planned, or has occurred in the past 18 months
5. Participation in any interventional study (investigational product or device) for treatment of achondroplasia or short stature
6. Has had bone-related surgery impacting assessment of anthropometric measurements or is expected to have it during the study period. Children with previous limb-lengthening surgery may enroll if surgery occurred at least 18 months prior to the date of consent/assent and healing is complete without sequelae as determined by the investigator
7. Has any condition that in the view of the investigator places the child at high risk of poor compliance with the visit schedule or of not completing the study.
8. Any concurrent disease or condition that in the view of the investigator would interfere with study participation

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: It is assumed that each of the study sites will enroll approximately 10-15 children of both genders and of various ages (0-10 years old).
  The total number of children planned to be enrolled across all sites is approximately 200.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (57):
- United States (14):
  - Los Angeles Biomedical Research Institute At Harbour-UCLA Medical Centre, Los Angeles, California
  - Los Angeles BioMedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Alfred I. duPont Hospital for Children - Wilmington, Wilmington, Delaware
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - The John Hopkins, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Boston Childrens Hospital, Boston, Massachusetts
  - Univesity of Missouri - Columbia, Columbia, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children Hospital, Houston, Texas
  - Texas Children'S Hospital, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Australia (2):
  - Murdoch Childrens Research Institute, Parkville, Victoria
  - Childrens Hospital Melbourne, Melbourne
- Belgium (2):
  - Antwerp University Hospital, Antwerp
  - Universitair Ziekenhuis Antwerpen (UZA), Edegem
- Canada (3):
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - The Hospital for Sick Children, Toronto
- China (2):
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Beijing Children's Hospital, Capital Medical University, Beijing
- Denmark (2):
  - Righospitalet, Copenhagen
  - Bispebjerg Hospital, Copenhagen
- France (3):
  - Centre Hospitalier Universitaire La Timone, Marseille
  - Centre Hospitalier Univesitaire La Timone, Marseille
  - Hopital Necker-Enfants Malades, Paris
- Germany (4):
  - Center for Rare Skeletal Diseases in Childhood and Adolescence, Cologne
  - University Hospital of Cologne, Cologne
  - Otto-von-Guericke- Universitat Magdeburg, Magdeburg
  - Otto-von-Guericke-Universitat Magdeburg, Magdeburg
- Italy (7):
  - ASST Lariana Como, San Fermo della Battaglia, COMO
  - IRCCS Istituto Giannina Gaslini, Genova, Genoa
  - ASST Lariana Como, Como
  - IRCCS Istituto Giannina Gaslini, Genova
  - San Raffaele Hospital, Milan
  - Center for Rare Diseases, Department of Pediatrics, Polo Salute Donna e Bambino, Rome
  - Fondazione Policlinico Universitario A.Gemelli, Rome
- Japan (3):
  - Osaka Women's and Children's Hospital, Izumi, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Okayama University Hospital, Okayama
- Portugal (2):
  - Hospital Pediatrico de Coimbra, Coimbra
  - Hospital Pediátrico de Coimbra, Coimbra
- Spain (3):
  - Vall d'Hebron University Hospital, Barcelona
  - Vall D'Hebron Univeristy Hospital, Barcelona
  - Hospital Quironsalud Malaga, Málaga
- Switzerland (2):
  - CENTRE HOSPITALIER UNIVERSITAIRE VAUDOIS -CHUV Hôpital Neslé, Lausanne
  - Centre Hospitalier Universitaire Vaudois -CHUV, Lausanne
- United Kingdom (8):
  - Bristol Royal Childrens Hospital, Bristol
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Guy's & St Thomas NHS Trust, St Thomas' Hospital, London
  - Guys & St Thomas NHS Trust, London
  - Newcastle Hospital NHS Foundation Trust, Newcastle
  - Newcastle Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Sheffield Children's NHS Foundation Trust, Sheffield
  - Sheffield Childrens NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=TA46-002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective, registry study, and conducted at multiple clinical centers globally. A total of 315 participants with eligibility-verified were enrolled.
Groups:
- Enrolled Participants: Participants with achondroplasia were followed over 4 years with respect to achondroplasia symptoms, tests and treatments, anthropometric parameters and biomarkers of bone growth. No study intervention was administered, and no other type of therapy was provided.
Period: Overall Study
Arm/Group | Enrolled Participants
Started | 315
Completed | 4
Not Completed | 311
Not completed — Other | 10
Not completed — Withdrawal by Subject | 66
Not completed — The child is enrolled in an interventional study | 70
Not completed — Inclusion/exclusion criteria | 8
Not completed — At sponsor's request | 151
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: Baseline population included all enrolled participants.
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 315
Age, Customized [Count of Participants; unit: Participants]
  0-2 Years | 82
  2-10 Years | 213
  ≥10 Years | 18
  Missing age | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137
  Male | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 288
  Unknown or Not Reported | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 52
  Black or African American | 2
  White | 233
  Other | 24
  Not Applicable | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Standing Height
Description: Standing height (for participants aged ≥2 years) is an assessment of maximum vertical size. Standing height was measured using a stadiometer with a fixed vertical backboard and an adjustable head piece. Height in supine position (or length for participants aged <2 years) was measured using measuring board. Three valid measurements were performed at each visit and the average of the 3 valid measurements was reported and used in descriptive summaries. Data is reported according to age group (<2 years and ≥2 years) and gender of the participants.
Time Frame: Baseline, 1 year, 2 years, 3 years, 4 years
Population: Analysis population included all enrolled participants, among whom, 2 participants have not been included due to missing age. The "Overall Number of Participants Analyzed" was based on age at baseline. The "Number Analyzed" in a row was based on actually analyzed participants at each visit.
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Groups:
- Male (Aged <2 Years); Female (Aged <2 Years); Male (Aged ≥2 Years); Female (Aged ≥2 Years): Participants with achondroplasia were followed over a five-year period with respect to achondroplasia symptoms, tests and treatments, anthropometric parameters and biomarkers of bone growth. No study intervention was administered, and no other type of therapy was provided.
Arm/Group | Male (Aged <2 Years) | Female (Aged <2 Years) | Male (Aged ≥2 Years) | Female (Aged ≥2 Years)
Number analyzed (Participants) | 45 | 37 | 131 | 100
centimeter (cm)
  Baseline: number analyzed (Participants) | 45 | 35 | 125 | 91
  Baseline | 64.1 (6.50) | 61.8 (5.27) | 90.7 (12.26) | 88.8 (11.52)
  Change at 1 year: number analyzed (Participants) | 15 | 13 | 82 | 59
  Change at 1 year | 8.4 (5.74) | 9.6 (2.53) | 4.6 (1.30) | 4.8 (1.44)
  Change at 2 years: number analyzed (Participants) | 2 | 3 | 49 | 42
  Change at 2 years | 18.8 (1.72) | 15.7 (4.94) | 8.8 (2.03) | 9.0 (2.01)
  Change at 3 years: number analyzed (Participants) | 0 | 0 | 30 | 18
  Change at 3 years |  |  | 12.5 (2.69) | 13.4 (2.79)
  Change at 4 years: number analyzed (Participants) | 0 | 0 | 2 | 0
  Change at 4 years |  |  | 11.6 (2.03) |

2. Primary Outcome: Change From Baseline in Sitting Height
Description: Sitting height (for participants aged ≥2 years) is a measure of the trunk of the body from the buttocks to the top of the head when the participant is sitting upright. Sitting height was measured using a stadiometer and sitting height table. Crown-rump length (for participants aged <2 years) was measured using measuring board. Three valid measurements were performed at each visit and the average of the 3 valid measurements was reported and used in descriptive summaries. Data is reported according to age group (<2 years and ≥2 years) and gender of the participants.
Time Frame: Baseline, 1 year, 2 years, 3 years, 4 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Male (Aged <2 Years) | Female (Aged <2 Years) | Male (Aged ≥2 Years) | Female (Aged ≥2 Years)
Number analyzed (Participants) | 45 | 37 | 131 | 100
cm
  Baseline: number analyzed (Participants) | 45 | 35 | 125 | 91
  Baseline | 46.2 (4.39) | 44.8 (3.54) | 61.3 (6.78) | 59.9 (6.64)
  Change at 1 year: number analyzed (Participants) | 15 | 13 | 81 | 59
  Change at 1 year | 7.5 (5.66) | 6.7 (1.49) | 2.6 (1.06) | 2.9 (1.11)
  Change at 2 years: number analyzed (Participants) | 2 | 3 | 49 | 42
  Change at 2 years | 14.3 (1.11) | 10.8 (3.41) | 4.9 (1.49) | 5.6 (1.27)
  Change at 3 years: number analyzed (Participants) | 0 | 0 | 29 | 18
  Change at 3 years |  |  | 7.0 (1.74) | 7.8 (1.85)
  Change at 4 years: number analyzed (Participants) | 0 | 0 | 2 | 0
  Change at 4 years |  |  | 6.3 (1.65) |

3. Primary Outcome: Change From Baseline in Knee Height
Description: Knee height means lower segment length (lower segment=standing height - sitting height). Knee height was measured using knee height caliper. Three valid measurements were performed at each visit and the average of the 3 valid measurements was reported and used in descriptive summaries. Data is reported according to age group (<2 years, 2-10 years, and ≥10 years) and gender of the participants.
Time Frame: Baseline, 1 year, 2 years, 3 years, 4 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Male (Aged 2-10 Years); Female (Aged 2-10 Years); Male (Aged ≥10 Years); Female (Aged ≥10 Years): Participants with achondroplasia were followed over a five-year period with respect to achondroplasia symptoms, tests and treatments, anthropometric parameters and biomarkers of bone growth. No study intervention was administered, and no other type of therapy was provided.
Arm/Group | Male (Aged <2 Years) | Female (Aged <2 Years) | Male (Aged 2-10 Years) | Female (Aged 2-10 Years) | Male (Aged ≥10 Years) | Female (Aged ≥10 Years)
Number analyzed (Participants) | 45 | 37 | 119 | 94 | 12 | 6
cm
  Baseline: number analyzed (Participants) | 43 | 35 | 119 | 93 | 12 | 6
  Baseline | 15.0 (2.16) | 14.0 (1.92) | 22.5 (3.91) | 21.9 (3.69) | 29.1 (3.64) | 27.8 (2.70)
  Change at 1 year: number analyzed (Participants) | 22 | 17 | 79 | 59 | 6 | 3
  Change at 1 year | 2.3 (1.39) | 2.7 (0.95) | 1.6 (1.00) | 1.5 (0.93) | 1.3 (0.83) | 1.4 (0.16)
  Change at 2 years: number analyzed (Participants) | 17 | 17 | 48 | 48 | 5 | 0
  Change at 2 years | 4.6 (1.03) | 4.8 (1.44) | 3.2 (1.96) | 3.4 (1.44) | 2.0 (0.41) |
  Change at 3 years: number analyzed (Participants) | 8 | 9 | 26 | 22 | 4 | 0
  Change at 3 years | 6.2 (0.95) | 6.4 (1.85) | 4.5 (2.31) | 5.0 (1.99) | 3.4 (0.99) |
  Change at 4 years: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0
  Change at 4 years |  |  | 3.5 (1.25) |  |  |

4. Primary Outcome: Change From Baseline in Head Circumference
Description: Head circumference is a measurement of the circumference of the child's head at its largest area, above the eyebrows and ears and around the back of the head. Head circumfernce was measured using measuring tape. Three valid measurements were performed at each visit and the average of the 3 valid measurements was reported and used in descriptive summaries. Data is reported according to age group (<2 years, 2-10 years, and ≥10 years) and gender of the participants.
Time Frame: Baseline, 1 year, 2 years, 3 years, 4 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Male (Aged <2 Years) | Female (Aged <2 Years) | Male (Aged 2-10 Years) | Female (Aged 2-10 Years) | Male (Aged ≥10 Years) | Female (Aged ≥10 Years)
Number analyzed (Participants) | 45 | 37 | 119 | 94 | 12 | 6
cm
  Baseline: number analyzed (Participants) | 45 | 37 | 119 | 93 | 12 | 6
  Baseline | 48.9 (3.75) | 47.7 (3.10) | 55.5 (2.28) | 54.4 (2.42) | 57.2 (2.56) | 55.2 (2.11)
  Change at 1 year: number analyzed (Participants) | 24 | 18 | 79 | 59 | 6 | 3
  Change at 1 year | 3.8 (2.31) | 4.0 (2.43) | 0.6 (0.70) | 0.4 (1.02) | 0.2 (0.43) | 0.9 (0.51)
  Change at 2 years: number analyzed (Participants) | 18 | 18 | 48 | 49 | 5 | 0
  Change at 2 years | 5.6 (3.27) | 5.3 (2.79) | 0.9 (0.74) | 1.1 (0.71) | 1.0 (0.38) |
  Change at 3 years: number analyzed (Participants) | 9 | 9 | 26 | 22 | 4 | 0
  Change at 3 years | 4.7 (2.22) | 4.6 (2.88) | 1.0 (0.70) | 1.4 (0.55) | -0.4 (3.68) |
  Change at 4 years: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0
  Change at 4 years |  |  | 1.1 (0.09) |  |  |

5. Primary Outcome: Change From Baseline in Arm Span
Description: Arm span measurement is the distance between fingertips when the arms are outstretched. All participants should be measured supine lying on the measurement grid. Three valid measurements were performed at each visit and the average of the 3 valid measurements was reported and used in descriptive summaries. Data is reported according to age group (<2 years, 2-10 years, and ≥10 years) and gender of the participants.
Time Frame: Baseline, 1 year, 2 years, 3 years, 4 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Male (Aged <2 Years) | Female (Aged <2 Years) | Male (Aged 2-10 Years) | Female (Aged 2-10 Years) | Male (Aged ≥10 Years) | Female (Aged ≥10 Years)
Number analyzed (Participants) | 45 | 37 | 119 | 94 | 12 | 6
cm
  Baseline: number analyzed (Participants) | 44 | 36 | 118 | 89 | 12 | 6
  Baseline | 56.5 (6.13) | 55.2 (5.89) | 80.5 (11.07) | 79.4 (11.51) | 99.3 (10.09) | 99.3 (3.54)
  Change at 1 year: number analyzed (Participants) | 23 | 18 | 78 | 55 | 6 | 3
  Change at 1 year | 7.7 (1.94) | 8.6 (2.02) | 4.2 (1.63) | 4.4 (1.76) | -1.1 (10.93) | 4.2 (1.16)
  Change at 2 years: number analyzed (Participants) | 17 | 17 | 46 | 45 | 5 | 0
  Change at 2 years | 12.8 (2.40) | 14.3 (3.16) | 8.6 (2.24) | 8.7 (2.41) | 7.2 (0.88) |
  Change at 3 years: number analyzed (Participants) | 9 | 9 | 26 | 20 | 4 | 0
  Change at 3 years | 17.0 (2.16) | 17.9 (4.29) | 11.6 (2.71) | 12.4 (2.69) | 10.7 (0.96) |
  Change at 4 years: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0
  Change at 4 years |  |  | 10.1 (2.19) |  |  |

6. Primary Outcome: Number of Participants With Achondroplasia-Related Treatments
Description: Achondroplasia-related treatments were collected in a prospective and standardized fashion to allow characterization of the natural history of the disease course in the youngest participants in relation to the level of actual disease burden over time due to treatments, as well as data to support identification of possible risk factors. Data is reported according to the gender of the participants.
Time Frame: Baseline to end of study visit (up to 55 months)
Population: Analysis population included all enrolled participants.
Measure: Count of Participants; unit: Participants
Groups:
- Male (All Ages); Female (All Ages): Participants with achondroplasia were followed over a five-year period with respect to achondroplasia symptoms, tests and treatments, anthropometric parameters and biomarkers of bone growth. No study intervention was administered, and no other type of therapy was provided.
Arm/Group | Male (All Ages) | Female (All Ages)
Number analyzed (Participants) | 178 | 137
Participants
  Ear Tube Insertion | 32 | 17
  Adenoidectomy | 26 | 7
  Physiotherapy | 21 | 11
  Decompressive Craniectomy | 11 | 11
  Speech Rehabilitation | 13 | 9
  Tonsillectomy | 13 | 4
  Adenotonsillectomy | 11 | 5
  Continuous Positive Airway Pressure | 7 | 3
  Spinal Support | 6 | 3
  Occupational Therapy | 5 | 2
  Oxygen Therapy | 3 | 4
  Myringotomy | 5 | 1
  Bilevel Positive Airway Pressure | 4 | 0
  Mechanical Ventilation | 3 | 1
  Specialist Consultation | 3 | 1
  Epiphysiodesis | 1 | 2
  Ergotherapy | 2 | 1
  Psychotherapy | 2 | 1
  Spinal Decompression | 2 | 1
  Bone Operation | 2 | 0
  Dental Care | 1 | 1
  Middle Ear Operation | 2 | 0
  Orthodontic Procedure | 1 | 1
  Spinal Laminectomy | 2 | 0
  Ventriculo-Peritoneal Shunt | 1 | 1
  Hearing Aid Therapy | 1 | 0
  Kinesitherapy | 0 | 1
  Laryngoplasty | 1 | 0
  Mastoidectomy | 1 | 0
  Maxillofacial Operation | 1 | 0
  Medical Device Removal | 1 | 0
  Nasal Irrigation | 0 | 1
  Nasal Operation | 0 | 1
  Orthopaedic Insoles | 1 | 0
  Osteopathic Treatment | 1 | 0
  Pharyngeal Operation | 1 | 0
  Pharyngeal Reconstruction | 1 | 0
  Posterior Fossa Decompression | 1 | 0
  Splint Application | 0 | 1
  Therapeutic Procedure | 0 | 1
  Tongue Tie Operation | 1 | 0
  Tooth Extraction | 1 | 0
  Weight Loss Diet | 1 | 0
  Magnetic Resonance Imaging | 3 | 3
  Audiogram | 3 | 2
  Magnetic Resonance Imaging Brain | 3 | 1
  Magnetic Resonance Imaging Neck | 2 | 1
  Magnetic Resonance Imaging Spinal | 2 | 1
  Sleep Study | 3 | 0
  Abdominal X-Ray | 1 | 0
  Acoustic Stimulation Tests Normal | 1 | 0
  Brain Stem Auditory Evoked Response | 1 | 0
  Bronchoscopy | 1 | 0
  Ear, Nose And Throat Examination | 1 | 0
  Electromyogram | 1 | 0
  Laryngoscopy | 1 | 0
  Neurological Examination Abnormal | 0 | 1
  Otoacoustic Emissions Test | 1 | 0
  Otoscopy | 1 | 0
  Skeletal Survey | 0 | 1
  Sleep Endoscopy | 1 | 0
  Somatosensory Evoked Potentials | 0 | 1
  Ultrasound Scan | 1 | 0
  Ultrasound Skull | 1 | 0
  Hearing Aid User | 3 | 1
  Walking Aid User | 1 | 0
  Cervical Spinal Stenosis | 0 | 1
  Kyphosis | 0 | 1
  Lordosis | 0 | 1
  Foramen Magnum Stenosis | 0 | 1
  Otitis Media Chronic | 0 | 1

7. Secondary Outcome: Baseline and Post-baseline Measurements of Serum Collagen X Marker
Description: Collagen X Marker (CXM), is a degradation by-product of endochondral ossification that is released into the circulation in proportion to overall growth plate activity. This marker corresponds to the rate of linear bone growth at time of measurement as recently demonstrated in children of normal average growth. Data is reported according to age group (<2 years, 2-10 years, and ≥10 years) and gender of the participants.
Time Frame: Baseline, 1 year, 2 years, 3 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per liter (ng/L)
Arm/Group | Male (Aged <2 Years) | Female (Aged <2 Years) | Male (Aged 2-10 Years) | Female (Aged 2-10 Years) | Male (Aged ≥10 Years) | Female (Aged ≥10 Years)
Number analyzed (Participants) | 45 | 37 | 119 | 94 | 12 | 6
nanogram per liter (ng/L)
  Baseline: number analyzed (Participants) | 35 | 27 | 101 | 77 | 12 | 6
  Baseline | 20433 (8479.2) | 20998 (8959.5) | 15336 (4360.7) | 15516 (5019.8) | 11798 (4330.0) | 14433 (2433.7)
  1 year: number analyzed (Participants) | 19 | 16 | 70 | 56 | 6 | 3
  1 year | 16053 (6025.0) | 18767 (5128.7) | 15623 (4208.9) | 15820 (4830.7) | 13815 (4726.9) | 13343 (4635.4)
  2 years: number analyzed (Participants) | 17 | 15 | 38 | 45 | 5 | 0
  2 years | 13757 (3906.2) | 17534 (5558.0) | 14046 (4520.1) | 15172 (4932.6) | 13630 (4404.8) |
  3 years: number analyzed (Participants) | 9 | 8 | 25 | 20 | 3 | 0
  3 years | 13719 (3198.7) | 14953 (3227.0) | 14416 (3943.9) | 14088 (4463.0) | 13597 (6226.5) |

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from screening to end of study visit (up to 55 months).
Description: An AE is defined as any untoward medical occurrence and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease, whether or not related to the participant's participation in the study. Any AE that occurred from the time the participant consented to the clinical research through and including 12 hours after completion of the qualifying procedure was recorded.
Arm/Group | Enrolled Participants
All-Cause Mortality (participants affected / at risk) | 0/315
Serious Adverse Events (participants affected / at risk) | 0/315
Other Adverse Events (participants affected / at risk) | 0/315

LIMITATIONS AND CAVEATS:
The study was early terminated due to lack of efficacy in the Phase 2 study. The observation period was less than the planned 5 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT03794609/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT03794609/SAP_001.pdf